CLINICAL TRIAL: NCT07075614
Title: The Effectiveness of a Parent Training Program for Children With Autism Spectrum Disorder and High-Risk Infants: A Case-Control Study
Acronym: PTP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Collaborators: Istanbul Instıtute of Child And Adolescent Psychiatry (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Canan Tanıdır, Prof Dr, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HRU.23.20.36
Record Dates: First submitted 2025-07-09; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Autism Disorder
Keywords: autism; parent training program
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Parent Training Program + Routine Care
  Interventions: Behavioral: Parent Training Program
- Control Group (No Intervention): Routine Care

INTERVENTIONS:
Behavioral: Parent Training Program — Parent Training Programs are complementary interventions to special education, implemented by parents to support the social, cognitive, and behavioral development of children with autism and other developmental disorders.
  Throughout the program, key developmental skills that children are expected to acquire-such as social skills (eye contact, joint attention, play, imitation), language, cognitive, motor, and self-care abilities-are explained using sample photos and simple instructions.
  Additionally, the program provides guidance on how to foster secure attachment between parent and child and how to support social-communicative skills through warm, responsive interactions in daily life.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to evaluate the effectiveness of a parent training program on the severity of autism-related symptoms in two groups: (1) infants under the age of 2 who show early signs of autism, and (2) children aged 2 to 5 years who have been diagnosed with Autism Spectrum Disorder (ASD). The study also aims to assess the program's impact on the quality of life and stress levels of the children's parents or caregivers.

The study will include children aged 0 to 5 years who are either considered at risk for autism or have an ASD diagnosis, along with their caregivers. A total of 250 participants are expected to enroll in the study. Informed consent will be obtained from all parents or caregivers before participation.

After consent, the 250 children will be randomly assigned to one of two groups:

Group A: Parent Training Program + Routine Care Group B: Routine Care Only While Group B will receive standard treatments such as education and psychotherapy and a single psychoeducational session about autism and its treatment, Group A will receive the same routine care plus the structured Parent Training Program.

Children in both groups will be assessed before the intervention begins and again after 12 weeks. Evaluations will be conducted with the support of professionals using standardized tools. Caregivers will complete a background information form with the help of the research team.

To assess symptom severity, the Modified Checklist for Autism in Toddlers (M-CHAT), the Childhood Autism Rating Scale (CARS), and the Clinical Global Impression Scale (CGI) will be administered by clinicians. General developmental levels will be evaluated using screening tools such as the Denver Developmental Screening Test or AGTE. Caregivers will also complete the Quality of Life in Autism-Parent Version and the Parenting Stress Index.

ELIGIBILITY:
Inclusion Criteria:

* Having a child over the age of 2 diagnosed with Autism Spectrum Disorder (ASD), or having a high-risk infant under the age of 2 showing signs of autism
* Willingness to participate in the study
* Parent/caregiver must have completed at least primary school education

Exclusion Criteria:

* Refusal to participate in the study
* The child has a sensory, physical, or neurological disorder
* The parent or primary caregiver has a diagnosed psychiatric disorder that significantly impairs functioning
* The parent or caregiver has any physical illness that affects their interaction with the child (e.g., physical disability, visual or auditorial impairment)

Ages: 0 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Autism Severity as Measured by the Childhood Autism Rating Scale (CARS) | Baseline, After 1 and 3 Months from Intervention
  Autism severity will be assessed using the Childhood Autism Rating Scale (CARS), a clinician-rated tool that evaluates behavior in 15 areas related to communication, social interaction, and sensory responses. Each item is rated on a scale from 1 (no signs of autism) to 4 (severe symptoms), with a total score ranging from 15 to 60.
  The total CARS score will be recorded at baseline (prior to intervention) and again.
  The primary outcome is the change in total score, which reflects improvement or worsening in the severity of autism symptoms over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No